CLINICAL TRIAL: NCT05125237
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM)- Amiloride vs Triamterene
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2019A010961-7
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amiloride; Triamterene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amiloride: Exposure group
  Interventions: Drug: Amiloride
- Triamterene: Reference group
  Interventions: Drug: Triamterene

INTERVENTIONS:
Drug: Amiloride — Amiloride claim is used as the exposure group.
  Groups: Amiloride
Drug: Triamterene — Triamterene claim is used as the reference group.
  Groups: Triamterene

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://docs.google.com/spreadsheets/d/1IdoLUI5-bz_1D_0IflZovJO9e1_3kFLc_JLEFM030No/edit?usp=sharing or Appendix A for full code and algorithm definitions.

Medicare timeframe: 2008 to 2018 (end of data availability).

Inclusion Criteria:

* 1. Aged > 65 years on the index date
* 2. Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date
* 3. At least two claims with hypertension diagnosis recorded in 365 days prior to cohort entry date

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. Prior use of amiloride or triamterene any time prior to cohort entry date

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will employ a new user, active comparator, observational cohort study design comparing amiloride to triamterene. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of amiloride or triamterene (index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).
Sampling Method: Non-Probability Sample
Enrollment: 155963 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amiloride | Triamterene
Started | 7476 | 148487
Completed | 7305 | 7305
Not Completed | 171 | 141182

BASELINE CHARACTERISTICS:
Population: Study cohort after 1:1 propensity score matching
Groups:
- Total: Total of all reporting groups
Arm/Group | Amiloride | Triamterene | Total
Number analyzed (Participants) | 7305 | 7305 | 14610
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 7305 | 7305 | 14610
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.06 (6.61) | 74.22 (6.77) | 74.14 (6.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4253 | 4219 | 8472
  Male | 3052 | 3086 | 6138
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6019 | 6054 | 12073
  Black | 825 | 782 | 1607
  Asian | 123 | 120 | 243
  Hispanic | 126 | 135 | 261
  Native American | 23 | 21 | 44
  Other | 124 | 124 | 248
  Unknown | 65 | 69 | 134
Dementia risk factors [Count of Participants; unit: Participants]
  Diabetes | 5784 | 5819 | 11603
  Obesity | 1979 | 1961 | 3940
  Coronary artery disease | 3087 | 3182 | 6269
  Depression | 1168 | 1130 | 2298
  Anxiety | 1104 | 1108 | 2212
  Bipolar disorder | 121 | 143 | 264
  Schizophrenia | 42 | 53 | 95

OUTCOME MEASURES:

1. Primary Outcome: Time to Dementia Onset
Description: Time to dementia onset, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition due to size limitations.
Time Frame: Median follow up times: 1) 119 days (exp), 111 days (ref) 2) 859 days (exp), 852 days (ref) 3) 333 days (exp), 286 days (ref) 4) 120 days (exp), 111 days (ref)
Population: Study cohort after 1:1 propensity score matching
Measure: Number (95% Confidence Interval); unit: Incidence rate per 1000 person year
Arm/Group | Amiloride | Triamterene
Number analyzed (Participants) | 7305 | 7305
Incidence rate per 1000 person year
  Analysis 1 | 12.6 [10.1 to 15.6] | 14.8 [11.9 to 18.2]
  Analysis 2 | 20.9 [17.5 to 24.8] | 21.5 [18.0 to 25.4]
  Analysis 3 | 12.2 [9.2 to 16.0] | 17.4 [13.6 to 21.9]
  Analysis 4 | 2.4 [1.4 to 3.8] | 4.3 [2.8 to 6.3]

ADVERSE EVENTS:
Time Frame: 'As-treated' follow-up approach - Median follow-up days of 119 (for Amiloride) and 111 (for Triamterene)
Description: Our study did not capture Serious Adverse Events.
Arm/Group | Amiloride | Triamterene
All-Cause Mortality (participants affected / at risk) | 0/7305 | 0/7305
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/7305 | 0/7305

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT05125237/Prot_SAP_002.pdf